CLINICAL TRIAL: NCT05979142
Title: A Prospective Cohort Study of a Community-based Primary Care Program's Effects on Pharmacotherapy Quality in Low-income Peruvians With Type 2 Diabetes and Hypertension
Brief Title: Community-based Primary Care Program Effects on Pharmacotherapy of Type 2 Diabetes and Hypertension in Peru
Status: Completed | Type: Observational
Sponsor: Asociación Siempre Salud (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1912252903
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: low and middle income countries; primary care; chronic care model; community health workers; cohort study; pharmacotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- program (pre-exposure): During the pre-exposure period, usual care was provided by two public hospitals, several Ministry of Health clinics, private clinics and pharmacies, and Siempre Salud.
- program (post-exposure): The program had components of four Chronic Care Model (CCM) elements (delivery system design, self-management, decision support, and community resources), community health workers (CHWs), and no out-of-pocket costs for visits and medications.
  Interventions: Other: community-based primary care program

INTERVENTIONS:
Other: community-based primary care program — See group description
  Groups: program (post-exposure)

SUMMARY:
The goal of this observational study is to compare usual care to a community-based primary care program (having components of treatment decisions based on clinical guidelines, self-management education, community health workers, and free health care visits and medications) in low-income Peruvians with type 2 diabetes and/or hypertension.

The main question[s] it aims to answer are:

* Compared to pre-program usual care, does the program result in greater benefits, measured as greater proportions of patients with glucose and blood pressure control or maximal quantities and doses of medications?
* Are there greater benefits when the program was provided at home compared to when the program was provided in a clinic?
* Does longer participation in the program result in greater benefits?

Participants will participate in:

* Self-management education provided by community health workers.
* Monitoring of healthy behaviors and glucose, blood pressure, and weight.
* Receipt of free medications for blood pressure, glucose, and heart disease prevention.

DETAILED DESCRIPTION:
A pre-post study of visit-level data gathered prospectively during a community-based primary care program evaluated its effects on pharmacotherapy of type 2 diabetes and hypertension. The program was conducted by Asociación Siempre Salud, a Peruvian non-profit organization, in three neighborhoods ("the community") in Pueblo Nuevo, Chincha District, Peru. Door-to-door surveys identified all persons residing in the study community. Persons > 35 years old were eligible, without exclusions, to participate in type 2 diabetes and hypertension screening and diagnosis. Most participated in mass screenings between September and December 2011, others in later ad hoc screenings. Patients with negative screening results on medications were re-screened following medication withdrawal. Those with confirmed diagnoses were eligible to participate in the program.

Three binary exposures were evaluated for their effects on adherence to four treatment standards and one composite standard: 1) 'program exposure' (post- vs. pre-exposure); 2) 'program retention in care' (>50% of allowable time in both home and clinic care periods, compared to <50% in either care period (but not both)), and 3) 'care period', (clinic compared to home care). 'Care period treatment time' (>50% of allowable time versus less) was evaluated as an independent variable in the study of the care period exposure.

During the pre-exposure period, usual care was provided by two public hospitals, several Ministry of Health clinics, private clinics and pharmacies, and Siempre Salud. The program, to which patients were then exposed, had components of four CCM elements (delivery system design, self-management, decision support, and community resources), CHWs, and no out-of-pocket costs for visits and medications. Self-management was based on national standards and utilized educational materials from professional societies and government agencies in the USA. Decision support consisted of guidelines-based standards adapted to our low-resource setting and simplified medication treatment protocols for diabetes, hypertension, and primary prevention of CVD. The delivery system consisted of two care models employed sequentially: first home care, then clinic care (see care period exposure).

During the home care period, the physician made an initial visit, after which CHWs made weekly visits to patients' homes. CHWs monitored clinical parameters, provided self-management education and support, tracked self-care behaviors, documented visits, acted on clinical alerts, and delivered medications. They entered encounter data into a spreadsheet and filled prescriptions under physician supervision. The physician made treatment decisions reliant on home visit data and patient care conferences. During the subsequent clinic period, patients made monthly visits to the clinic physician who provided all care.

ELIGIBILITY:
Inclusion Criteria:

35 years or older with confirmed diagnosis of type 2 diabetes and/or hypertension

Exclusion Criteria:

None

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three neighborhoods ("the community") in Pueblo Nuevo, Chincha District, Ica, Peru participated in the study. Peru is a middle-income country, but most people in the study community live below the poverty line. Door-to-door surveys identified all persons residing in the study community. Patients 35 years and older were eligible to participate in diabetes and hypertension screening. 83% of all eligible persons participated in mass screenings between September and December 2011. Others participated in later ad hoc screenings. Those with confirmed diagnoses of type 2 diabetes and/or hypertension were eligible to participate in the program.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic agent standard | 27 months
  Standard was defined as glycemic control or maximum doses of two hypoglycemic agents (metformin and glibenclamide) in eligible patients with type 2 diabetes.
Antihypertensive agent standard | 27 months
  Standard was defined blood pressure control or maximum doses of three or more antihypertensive agents in eligible patients with elevated blood pressure (>130/80 mm Hg in diabetics, >140/90 mm Hg in non-diabetics)
Angiotensin-converting enzyme inhibitor (ACEi) standard | 27 months
  Standard was defined as any ACEi in eligible patients with diabetes and elevated BP (>130/80 mm Hg).
Low-dose aspirin standard | 27 months
  Standard was defined as any low-dose aspirin in eligible patients with 10-year cardiovascular disease (CVD) risk >10%.
Composite standard | 27 months
  Coded 'yes' if all treatment standards for which eligible were achieved.

CONTACTS AND LOCATIONS:
Overall Officials: John E Deaver, MD, Principal Investigator — Asociación Siempre Salud

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data in the following formats: Stata (*.dta) and comma-delimited text (*.csv) files and a data dictionary will be shared with Dryad data repository.
Time Frame: during submission of manuscript for publication